CLINICAL TRIAL: NCT01806610
Title: A Randomized, Placebo-controlled Trial of BPS804 on Safety and Tolerability in Patients With Late-stage Chronic Kidney Disease
Brief Title: Study of Safety and Tolerability of BPS804 in Patients With Late-stage Chronic Kidney Disease
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Ultragenyx Pharmaceutical Inc (Industry)
Collaborators: Mereo BioPharma (Industry); Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CBPS804A2204; 2012-003348-63 (EudraCT Number)
Record Dates: First submitted 2013-03-03; First posted 2013-03-07 (Estimated); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Chronic-kidney Disease Stage 5D on Stable Hemodialysis
Keywords: Randomized; Placebo-controlled trial; BPS804; Safety, tolerability, and PK; Patients with late-stage chronic kidney disease.
MeSH Terms: interventions — setrusumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- BPS804 (Experimental): Single dose BPS804 administration.
  Interventions: Drug: BPS804
- Placebo (Placebo Comparator): Single dose placebo administration.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BPS804 — Single dose BPS804 administration.
  Other Names: Active BPS804.
  Arms: BPS804
Drug: Placebo — Single dose placebo administration.
  Other Names: BPS804 placebo.
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the safety, tolerability, and PK following a single administration of BPS804 in patients with chronic kidney disease stage 5D (CKD-5D) on hemodialysis.

DETAILED DESCRIPTION:
This study was previously posted by Novartis and was transferred to Ultragenyx in February 2021.

ELIGIBILITY:
Inclusion criteria

* Written informed consent must be obtained before any assessment is performed.
* Males and females aged 18 to 80 years included, with CKD-5D (GFR < 15 mL/min per 1.73m2) on stable hemodialysis as evidenced by monthly Kt/Vurea ≥ 1.20 (obtained from local laboratory) or urea reduction ratio ≥ 60% (obtained from local laboratory) for past 3 consecutive months prior to screening.
* Patient must be on maintenance renal replacement therapy (i.e., exclusively on standard hemodialysis with non-porous membrane) 3 times per week, for > 3 months before screening with a stable dialysis prescription, as defined by no change in material (i.e., dialyzer, filter/ membrane) type and dialysis duration for ≥ 4 weeks before screening.
* If patient is currently being treated with calcimimetics, the prescribed dose must be constant for at least 30 days prior to screening and should remain constant during the study duration.
* If patient is currently being treated with vitamin D, the prescribed dose must be constant for at least 30 days prior to screening and should remain constant during the study duration.
* Screening body mass index (BMI) between >18.5 and ≤ 35 kg/m2 and weigh of at least 50 kg.
* Able to communicate well with the investigator, to understand and comply with the requirements of the study.

Exclusion Criteria

* Patients who are on peritoneal dialysis.
* Patients who had a parathyroidectomy within 3 months prior to screening or patients who have a parathyroidectomy scheduled during the course of the study.
* Patients who have a kidney transplant scheduled during the study.
* Patients with clinically symptomatic spinal stenosis.
* Women who are pregnant or nursing (lactating).
* Women of child-bearing potential who are planning a pregnancy during the course and duration of the study.
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, must use highly effective contraception during the study and for 5 half-lives (i.e., around 10 weeks) after stopping treatment. Highly effective contraception is defined as either:

  1. Total abstinence: When this is in line with the preferred and usual lifestyle of the patient. [Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception].
  2. Sterilization: have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
  3. Male partner sterilization (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate). [For female study patients, the vasectomised male partner should be the sole partner for that patient].
  4. Use of a combination of any two of the following (1+2 or 1+3 or 2+3):

     1. Use of oral, injected or implanted hormonal methods of contraception.
     2. Placement of an intrauterine device (IUD) or intrauterine system (IUS).
     3. Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository.

In case of use of oral contraception women should have been stable on the same pill for a minimum of 3 months before taking study treatment.

* Liver disease or liver injury as indicated by abnormal liver function tests such as SGOT (AST), SGPT (ALT), γ-GT.
* Hemoglobin of ≤ 9 g/dL in male, and ≤ 8 g/dL in female patients. (Note: Treatment with erythropoietin-stimulating agents (ESA) is allowed).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-08; Primary Completion 2014-04 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Occurrence of adverse events after a single administration of BPS804 | 17 weeks
  Adverse events will be counted within each treatment and study part. The numbers and percentages of adverse events will be tabulated by body system, preferred term, and severity.

SECONDARY OUTCOMES:
Pharmacokinetic (PK) of BPS804 in serum: area under the serum concentration-time curve from time zero to the time of the last quantifiable concentration | Pre-dose, and 2, 24, 44, 48, 168 hours and 15, 22, 29, 57, and 85 days after dosing
  AUClast: The area under the serum concentration-time curve from time zero to the time of the last quantifiable concentration
PK of BPS804 in serum: area under the serum concentration-time curve from time zero to infinity | Pre-dose, and 2, 24, 44, 48, 168 hours and 15, 22, 29, 57, and 85 days after dosing
  AUCinf: The area under the serum concentration-time curve from time zero to infinity
PK of BPS804 in serum: observed maximum serum concentration following drug administration | Pre-dose, and 2, 24, 44, 48, 168 hours and 15, 22, 29, 57, and 85 days after dosing
  Cmax: The observed maximum serum concentration following drug administration
PK of BPS804 in serum: terminal elimination half-life | Pre-dose, and 2, 24, 44, 48, 168 hours and 15, 22, 29, 57, and 85 days after dosing
  T1/2: The terminal elimination half-life
PK of BPS804 in serum: time to reach the maximum concentration after drug administration | Pre-dose, and 2, 24, 44, 48, 168 hours and 15, 22, 29, 57, and 85 days after dosing
  Tmax: The time to reach the maximum concentration after drug administration
Concentration of BPS804 in dialysate 48 hours after dosing | Day 3, 48 hours post dosing
  Quantify BPS804 in dialysate 48 hours after dosing to assess any impact of dialysis on BPS804

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Ultragenyx Pharmaceutical Inc